CLINICAL TRIAL: NCT06484179
Title: Enhancing Motivation to Quit Smoking Via Self-Help Intervention Targeted to Cancer Type: A Pilot Randomized Control Trial (RCT)
Brief Title: Enhancing Motivation to Quit Smoking Via Self-Help Intervention Targeted to Cancer Type
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCI173619; K22CA276255-01 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Smoking
MeSH Terms: conditions — Neoplasms; Smoking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to (1) Usual Care or (2) Usual Care + targeted self-help intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care
- Usual Care + Targeted Self-Help Intervention (Experimental)
  Interventions: Behavioral: Targeted Self-Help

INTERVENTIONS:
Behavioral: Targeted Self-Help — In addition to usual care participants will receive a self-help booklet specific for their cancer type. There are five booklets available, written at a 5-6th grade reading level and targeted by cancer type, that explain the connection between smoking and each cancer type, describe the benefits of quitting smoking after cancer, and address some of the barriers cancer patients face to quit smoking when fighting cancer. Each booklet also includes four testimonials inspired from conversations with patients.
  Arms: Usual Care + Targeted Self-Help Intervention
Behavioral: Usual Care — Participants will receive the standard care typically offered for smoking cessation.
  Arms: Usual Care

SUMMARY:
The purpose of this research study is assess feasibility and acceptability of a recently developed brief self-help intervention targeted by cancer type to increase motivation to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who smoke and recently (i.e., within 6 months) received a diagnosis of breast, colorectal, gynecological, skin melanoma, or bladder cancer (n = 20 per cancer type). (Investigators will consider smokers individuals who report having smoked ≥1 cigarette in the past 30 days.)
* Able to read/write English;
* Able to give informed consent;
* Not currently enrolled in a smoking cessation program;
* Age ≥18 years old.

Exclusion Criteria:

* Male patients diagnosed with breast cancer will be excluded as lifetime risk for breast cancer in men is far below 1%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Number of participants who consent to participate in the study
Retention- Completion of 2-week follow-up | 2 weeks post-randomization
  Number of participants who complete the 2-week follow-up assessment
Retention- Completion of 1 month follow-up | 1 month post-randomization
  Number of participants who complete the 1 month follow-up assessment
Adherence- 2 weeks post-randomization | 2 weeks post-randomization
  Number of participants who read the booklet 2 weeks post-randomization
Adherence- 1 month post-randomization | 1 month post-randomization
  Number of participants who read the booklet 1 month post-randomization
Acceptability | 2 weeks post-randomization, 1 month post-randomization
  Treatment satisfaction measured with 8 items adapted from the Client Satisfaction Questionnaire. Values between 8 and 32 with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Motivation to quit smoking | Baseline, 2 weeks post-randomization, 1 month post-randomization
  Changes in motivation to quit smoking will be assessed using the Contemplation Ladder. This is a validated measure for the assessment of readiness to quit smoking on a scale from 0 to 10. Higher scores indicate greater motivation to quit smoking.
Treatment Engagement defined by the number of participants who enroll with the state tobacco quitline | 2 weeks post-randomization, 1 month post-randomization
  Engagement in smoking cessation services defined by enrollment with state tobacco quitline
Smoking Status | 2 weeks post-randomization, 1 month post-randomization]
  7-day point prevalence smoking abstinence (i.e., not smoking, not even a puff, in the past 7 days)
Smoking Status | 2 weeks post-randomization, 1 month post-randomization
  30-day point prevalence smoking abstinence (i.e., not smoking, not even a puff, in the past 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Martinez, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No